CLINICAL TRIAL: NCT02008461
Title: Botulinum Toxin Injection for Preventing Secondary Atrial Fibrillation in Patient With Supra-ventricular Tachyarrythmias
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BT_SVT
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Supra-ventricular Tachyarrhythmias
MeSH Terms: interventions — Radiofrequency Ablation; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RFA (Active Comparator): Mapping and radiofrequency ablation are performed by using standard methods.
  Interventions: Procedure: radiofrequency ablation
- RFA+BT injection (Active Comparator): Mapping and radiofrequency ablation are performed by using standard methods.
  Injection of the botulinum toxin is performed in main anatomical zones of ganglionated plexuses of left atrium using Myostar catheter (Biosense Webster).
  Interventions: Procedure: radiofrequency ablation; Drug: botulinum toxin injection

INTERVENTIONS:
Procedure: radiofrequency ablation
Drug: botulinum toxin injection
  Arms: RFA+BT injection

SUMMARY:
The investigators have conducted a prospective, double-blind, randomized study to assess the comparative safety and efficacy of two different ablation strategies, RFA versus RFA plus botulinum toxin injection, in patients with supra-ventricular tachyarrhythmias. Results were assessed with the use of an implanted monitoring device (IMD).

ELIGIBILITY:
Inclusion Criteria:

* atrial flutter, AV nodal re-entry tachycardia, focal atrial tachycardia, WPW syndrome
* secondary atrial fibrillation

Exclusion Criteria:

* congestive heart failure
* LV ejection fraction < 35%
* left atrial diameter > 60 mm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
number of episodes of atrial fibrillation | 1 year

SECONDARY OUTCOMES:
serious adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- University of Rochester, Rochester, New York, United States
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru